CLINICAL TRIAL: NCT03626350
Title: Prospective Evaluation of the Efficacy and Safety of Submucosal Endoscopy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0046
Record Dates: First submitted 2018-08-02; First posted 2018-08-13 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Neoplasia; Hirschsprung's Disease; Esophageal Obstruction; Gastroparesis; Spastic Esophageal Disorders; Zenker's Diverticulum
MeSH Terms: conditions — Hirschsprung Disease; Airway Obstruction; Gastroparesis; Zenker Diverticulum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To test the idea that submucosal endoscopy is effective and safe for endoscopic myotomy, endoscopic submucosal dissection, and access for tissue acquisition and resection. Submucosal endoscopy is a recent innovative addition to gastrointestinal endoscopy. This involves endoscopic maneuvers in the gut wall, by dissection of the submucosal layer of GI tract, thereby allowing endoscopic myotomy (incision of the muscle), endoscopic access for tissue acquisition and therapy, and resection of precancerous and cancerous gastrointestinal tissue. This approach has been a dramatic game-changer for minimally invasive management of various gastrointestinal conditions such as Zenker's diverticulum, Achalasia, Spastic Esophageal Disorders, Gastroparesis, esophageal obstruction, Hirschsprung's Disease, and Gastrointestinal neoplasia.

The aim of the proposed study is to prospectively assess technical success, clinical success, and adverse events after submucosal endoscopy. Technical success will be defined as ability to successfully complete the submucosal endoscopic procedure. Clinical success will be defined as symptom relief and objective evaluation which will be assessed with radiologic imaging, repeat endoscopy, gastrointestinal motility studies, and pathology results routinely performed post-procedure for clinical care, as indicated. Adverse events will be recorded per published ASGE criteria.

A database/ registry of patients undergoing submucosal endoscopic procedures will be created to demonstrate this.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo submucosal endoscopy
2. Age >18 years

Exclusion Criteria:

1. Age <18 years
2. Pregnancy
3. Coagulopathy (platelets less than 50, INR more than 1.8)

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A prospective database/registry of patients undergoing submucosal endoscopic procedures will be formed. Women and minorities will be included as they are frequently found to have indications for which submucosal endoscopic procedures may be indicated.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Technical and clinical success in performing submucosal endoscopy | baseline to one year
  Improvement in symptoms and objectively assessed by radiologic imaging, repeat endoscopy, gastrointestinal motility studies, and pathology.
Adverse Events | baseline to one year
  as defined by published ASGE criteria

SECONDARY OUTCOMES:
Procedure time | During procedure
  Procedure time
Submucosal endoscopy technique and device used | During procedure
  Submucosal endoscopy technique and device used

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States